CLINICAL TRIAL: NCT05510037
Title: Incidence and Prognostic Significance of HER-2 Status Discordance Between Primary Breast Cancer and Paired Recurrent/Metastatic Lesions
Status: Completed | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Jian Zhang,MD, Director of the phase I clinical trial department, Fudan University
Other Study IDs: YBCSG-22-08
Record Dates: First submitted 2022-08-15; First posted 2022-08-22 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- HER2-0
  Interventions: Other: no intervention
- HER2-LOW
  Interventions: Other: no intervention
- HER2-POSITIVE
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention was needed

SUMMARY:
About a half of HER2-negative breast cancer show HER2-low expression that can be targeted by new antibody-drug conjugates. The main aim of this study is to describe the evolution of HER2 expression from primary BC to relapse by including HER2-low category in both primary and recurrent BC samples. Patients with matched primary and relapse BC samples were included. 1299 patients were included.

ELIGIBILITY:
Inclusion Criteria:

Patients with available HER2 status of primary breast cancer and relapse/metastases

Exclusion Criteria:

Patients with other malignancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with available HER2 status of primary breast cancer and relapse/metastases
Sampling Method: Probability Sample
Enrollment: 1299 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
overall survival | up to 200 months
  The overall survival (OS) was defined as time from the date of initial diagnosis of recurrent/metastatic disease to the date of death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Jian Zhang, PHD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No